CLINICAL TRIAL: NCT04192084
Title: Microvascular Partial Toe Transfer for Reconstruction of Traumatic Amputations of the Digits
Brief Title: Microvascular Partial Toe Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yousif Tarek El-Gammal, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Toe Transfer
Record Dates: First submitted 2019-11-29; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Amputation, Traumatic; Hand Injuries
MeSH Terms: conditions — Amputation, Traumatic; Hand Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Traumatic amputations of the digits (Experimental): we will perform microvascular partial toe transfer for patients with traumatic amputations of one or more digits
  Interventions: Procedure: microvascular partial toe transfer

INTERVENTIONS:
Procedure: microvascular partial toe transfer — we will perform microvascular partial toe transfer for patients with traumatic amputation of one or more digits

SUMMARY:
Microvascular partial toe transfer for reconstruction of traumatic amputation of the digits

DETAILED DESCRIPTION:
Microsurgical toe transfer has become a gold standard option for amputated digit reconstruction. It can be used to correct almost any thumb defect. However, for optimal functional and esthetic results, proper initial care, preoperative planning, proper selection of suitable techniques, adjunct or secondary procedures and proper, postoperative rehabilitation are important.

The transfer of a toe to replace an amputated thumb represents one of the first applications of microsurgical techniques, yet to this day remains an epitome of reconstructive surgery, restoring critical function and form to the hand-injured patient. While techniques have greatly evolved to permit the treatment of multiple finger amputations, dystrophic nails and pulps, and traumatized or arthritic joint, the amputated thumb retains its status among the most indubitable indications for toe transfer. Microsurgical techniques have been refined to such a degree that almost any ablative deformity of the thumb could be corrected with some form of toe transfer. The question, therefore, is not if a defect could be reconstructed, but whether the patient is willing to undergo reconstruction. The concepts of "adequate function" and "optimal function" are therefore of central importance when discussing treatment options with a patient. Obviously, these parameters will be different for each patient depending upon his/her vocation, avocations, and desires. For many people, adequate function might be expected with an amputation that retains some length of the proximal phalanx (assuming sufficient soft tissue coverage is present or can be provided). However, for patients who require full length of their thumb, or who desire optimal rather than adequate function, toe transfer should be considered.

At present, the decision to use a particular toe transfer technique is mostly based on the surgeon's preference and training. The current data are inadequate to make any comments with regards to donor site morbidity. Till such data are available, an evidence-based recommendation for the superiority of a specific type of toe-to-thumb transfer cannot be made. We hypothesis that partial toe transfer provides the best aesthetic and functional reconstruction and the least donor site morbidity amongst all other types of transfers.

ELIGIBILITY:
Inclusion Criteria:

* Patient from 18-50 years old
* one or more finger amputations
* Minimum follow-up period of 6 months

Exclusion Criteria:

* patients whose loss was due to congenital anomaly.
* Patients who did not have a minimum follow-up period of six months .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
short-term functional outcome | six months
  Using DASH (The Disabilities of the Arm, Shoulder and Hand) score Reference for Score: Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG) Am J Ind Med. 1996 Jun;29(6):602-8. Erratum in: Am J Ind Med 1996 Sep;30(3):372.
  The Institute for Work & Health are the copyright owners of the DASH and QuickDASH Outcome Measures (http://www.dash.iwh.on.ca/)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buncke HJ Jr, Buncke CM, Schulz WP. Immediate Nicoladoni procedure in the Rhesus monkey, or hallux-to-hand transplantation, utilising microminiature vascular anastomoses. Br J Plast Surg. 1966 Oct;19(4):332-7. doi: 10.1016/s0007-1226(66)80075-9. No abstract available. PMID 4959061
- [Background] Cobbett JR. Free digital transfer. Report of a case of transfer of a great toe to replace an amputated thumb. J Bone Joint Surg Br. 1969 Nov;51(4):677-9. No abstract available. PMID 5371970
- [Background] Wei FC, Chen HC, Chuang CC, Noordhoff MS. Simultaneous multiple toe transfers in hand reconstruction. Plast Reconstr Surg. 1988 Mar;81(3):366-77. doi: 10.1097/00006534-198803000-00009. PMID 3340671
- [Background] Wei FC, Lutz BS, Cheng SL, Chuang DC. Reconstruction of bilateral metacarpal hands with multiple-toe transplantations. Plast Reconstr Surg. 1999 Nov;104(6):1698-704. doi: 10.1097/00006534-199911000-00013. PMID 10541171
- [Background] Koshima I, Soeda S, Takase T, Yamasaki M. Free vascularized nail grafts. J Hand Surg Am. 1988 Jan;13(1):29-32. doi: 10.1016/0363-5023(88)90194-3. PMID 3351225
- [Background] Logan A, Elliot D, Foucher G. Free toe pulp transfer to restore traumatic digital pulp loss. Br J Plast Surg. 1985 Oct;38(4):497-500. doi: 10.1016/0007-1226(85)90007-4. PMID 4052709
- [Background] Wei FC, Chen HC, Chuang DC, Chen S, Noordhoff MS. Second toe wrap-around flap. Plast Reconstr Surg. 1991 Nov;88(5):837-43. doi: 10.1097/00006534-199111000-00016. PMID 1924570
- [Background] Chen SH, Wei FC, Chen HC, Hentz VR, Chuang DC, Yeh MC. Vascularized toe joint transfer to the hand. Plast Reconstr Surg. 1996 Dec;98(7):1275-84. doi: 10.1097/00006534-199612000-00025. PMID 8942916
- [Background] Lutz BS, Wei FC. Basic principles on toe-to-hand transplantation. Chang Gung Med J. 2002 Sep;25(9):568-76. PMID 12479617
- [Background] Lin PY, Sebastin SJ, Ono S, Bellfi LT, Chang KW, Chung KC. A systematic review of outcomes of toe-to-thumb transfers for isolated traumatic thumb amputation. Hand (N Y). 2011 Sep;6(3):235-43. doi: 10.1007/s11552-011-9340-x. Epub 2011 May 26. PMID 22942845
- [Background] Wei FC. Tissue preservation in hand injury: the first step to toe-to-hand transplantation. Plast Reconstr Surg. 1998 Dec;102(7):2497-501. doi: 10.1097/00006534-199812000-00039. PMID 9858192
- [Background] Yim KK, Wei FC. Intraosseous wiring in toe-to-hand transplantation. Ann Plast Surg. 1995 Jul;35(1):66-9. doi: 10.1097/00000637-199507000-00013. PMID 7574290
- [Background] Wilson CS, Buncke HJ, Alpert BS, Gordon L. Composite metacarpophalangeal joint reconstruction in great toe-to-hand free tissue transfers. J Hand Surg Am. 1984 Sep;9(5):645-9. doi: 10.1016/s0363-5023(84)80004-0. PMID 6386954
- [Background] Morrison WA, O'Brien BM, MacLeod AM. Thumb reconstruction with a free neurovascular wrap-around flap from the big toe. J Hand Surg Am. 1980 Nov;5(6):575-83. doi: 10.1016/s0363-5023(80)80110-9. PMID 7000885
- [Background] Wei FC, Chen HC, Chuang DC, Jeng SF, Lin CH. Aesthetic refinements in toe-to-hand transfer surgery. Plast Reconstr Surg. 1996 Sep;98(3):485-90. doi: 10.1097/00006534-199609000-00019. PMID 8700986